CLINICAL TRIAL: NCT06339346
Title: Analysis of Histopathological Factors Predictive of Lymph Node Involvement and Management Practices in pT1 Colorectal Cancers Treated by Primary Endoscopic Resection: a Retrospective Population-based Study
Brief Title: Analysis of Histopathological Factors Predictive of Lymph Node Involvement and Management Practices in pT1 Colorectal Cancers Treated by Primary Endoscopic Resection
Acronym: PROMOT1
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0028 - PROMOT1
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Colorectal Adenocarcinoma
Keywords: colorectal cancer; pathological risk factors
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancers (CRC) extending beyond the muscularis mucosae and invading the submucosa without extending beyond it are classified as pT1.

Among these, a number of lesions presenting pejorative criteria, notably histopathological, have a significant risk of lymph node invasion, and are therefore candidates for partial colectomy with lymph node dissection. Tumors deemed to be at low risk of lymph node involvement can be treated by endoscopy alone.

It should be noted that further surgical intervention is not without comorbid consequences, and that a significant proportion of post-surgical surgical specimens are free of cancerous lesions.

The aim of this study is therefore to analyze the current histopathological criteria predictive of lymph node invasion, in order to more accurately select candidates for surgical management.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with pT1 colorectal cancer (of adenocarcinoma subtype only) diagnosed from January the 1st, 2009 to December the 31st, 2020, with first endoscopic resection, in the area of Finistère (France)

Exclusion Criteria:

* other than adenocarcinoma
* other than T1
* primary surgical management
* neoadjuvant treatment
* refusal to data collection

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: pT1 colorectal cancer (of adenocarcinoma subtype only) diagnosed from January the 1st, 2009 to December the 31st, 2020, with first endoscopic resection, in the area of Finistère (France)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of lymph node invasion rates as a function of tumor characteristics | 10 years

SECONDARY OUTCOMES:
Population demographics | 10 years
lesion characteristics | 10 years
management | 10 years
recurrence | 10 years
survival | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement